CLINICAL TRIAL: NCT00137865
Title: A Phase 1, Open Label, Dose Escalation Study of the Safety, Tolerability and Preliminary Efficacy of Intraperitoneal EGEN-001 in Patients With Recurrent Epithelial Ovarian Cancer
Brief Title: Safety Study of phIL-12-005/PPC to Treat Recurrent Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decided to terminate the study early so they could begin a second dose-escalation study of EGEN-001 in combination with standard chemotherapy.
Sponsor: EGEN, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGEN-001-101
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — GEN-1

ARMS (1):
- EGEN-001 (Experimental)
  Interventions: Genetic: EGEN-001 (phIL-12-005/PPC)

INTERVENTIONS:
Genetic: EGEN-001 (phIL-12-005/PPC)

SUMMARY:
Ovarian cancer may be caused by a build-up of genetic defects, or damaged genes within the cells of the body. Because the genes are damaged, the body is unable to produce a group of proteins called cytokines which are used by the immune system to fight cancer and some infections. The investigational gene transfer agent EGEN-001 (phIL-12-005/PPC) contains the human gene for interleukin-12 [IL-12] (a cytokine) in a special carrier system designed to enter the cells and help the body produce cytokines.

This study has two purposes; the first is to determine what different strengths of EGEN-001 can be given safely without major side effects, and the second is to see if EGEN-001 is able to slow down the growth of ovarian cancer.

DETAILED DESCRIPTION:
EGEN-001-101 is a Phase 1, open label, non-randomized, dose escalation study in up to 18 (eighteen) patients (three to six patients in each of the first three cohorts, and up to nine patients in a fourth cohort or MTD). The fourth cohort (or MTD, if earlier) will be expanded in increments of three patients until a total of 18 patients have been enrolled.

Each patient will provide written dated informed consent prior to undergoing eligibility screening for entry into the study. Screening evaluations will be performed within 21 days prior to scheduled study drug administration. If all eligibility criteria are met, the patient will be enrolled and will be scheduled for placement of the IP catheter at least 7 days prior to the scheduled dosing (Day -7) to allow adequate time for healing around the catheter insertion site. Baseline evaluations will be performed prior to dosing. At that time the investigator will ensure that the patient remains eligible for participation.

All study drug will be administered on an inpatient basis and the patient will remain confined for 24 hours following study drug administration for evaluation of safety and collection of specified body fluid samples for plasmid IL-12-DNA and cytokine determinations. Each patient will receive the same dose of EGEN-001 once weekly for four weeks (administered on Day 0, Day 7, Day 14, and Day 21). Patients will undergo safety evaluations 1, 4 and 24 hours and 3 days following each dose. Patients will return to the clinic for safety evaluations three days, one week and five weeks (± one week) following the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Female and at least 19 years of age (or minimum legal age and competency to provide voluntary written informed consent for study participation)
* Have received previous treatment for ovarian cancer that included a platinum based chemotherapy regimen
* Have recurrent epithelial ovarian cancer
* Have a measurable tumor by computed tomography (CT) scan according to Response Evaluation Criteria in Solid Tumors (RECIST)
* Have an ECOG performance status score of 0, 1, or 2
* If of childbearing potential, agree to follow an acceptable method of birth control (e.g., abstinence, intrauterine device [IUD] or barrier method), as determined by the investigator, for the duration of the study. Hormonal contraceptives should not be used as the sole method of birth control.
* Have normal organ and marrow function as defined below:

  * Leukocytes ≥ 3,000/µL;
  * Absolute neutrophil count ≥ 1,500/µL;
  * Platelets ≥ 100,000/µL;
  * Total bilirubin within institutional limits;
  * SGOT/SGPT ≤ 2.5 X institutional upper limit of normal (ULN);
  * Creatinine within institutional normal limits; OR creatinine clearance ≥ 60mL/min/1.73m2 for patients with creatinine levels above institutional normal.
* Have electrocardiogram (ECG) without clinically significant abnormality, as determined by a qualified cardiologist
* Have the capability (caregiver) of performing IP site care while at home

Exclusion Criteria:

* A serious uncontrolled intercurrent medical illness or disorder including, but not limited to, ongoing or active infection, abdominal surgery, autoimmune disorders, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations which would limit compliance with study requirements
* Intraabdominal disease > 5 (five) centimeters in diameter
* Previous treatment with whole abdominal irradiation
* Intestinal dysfunction or suspected extensive adhesions from prior history or findings at laparoscopy
* Intrahepatic disease
* Any condition/anomaly that would interfere with the appropriate placement of the IP catheter for study drug administration
* Received investigational agents within three months prior to study drug dosing
* Receipt of any medications (in particular, systemic or topical steroids) or substances known to affect, or with the potential to affect, the activity of EGEN-001
* Life expectancy of less than three months
* Known human immunodeficiency virus (HIV) infection
* Positive HbsAg
* Positive hepatitis C virus (HCV) serology
* Prior IP drug administration
* Prior immunotherapy for ovarian cancer
* Chemotherapy within four weeks prior to placement of IP catheter
* Radiotherapy within eight weeks prior to placement of IP catheter
* Contraindication (either allergy or impaired renal function) to injection with contrast media for adequate evaluation of tumor size by CT scan
* Pregnant or breast feeding an infant

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-08; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and to assess the spectrum of toxicities of EGEN-001 when administered by intraperitoneal (IP) infusion in patients with recurrent epithelial ovarian cancer

SECONDARY OUTCOMES:
To assess the preliminary efficacy of EGEN-001 by monitoring detectable tumor burden in patients with recurrent epithelial cancer
To assess EGEN-001 distribution by measuring human interleukin-12 plasmid (phIL-12) DNA copy number in the blood and peritoneal fluid
To assess the biological effects of EGEN-001 on cytokine production by measuring interferon (IFN) gamma and interleukin-12 (IL-12) concentrations in the blood and peritoneal fluid

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Alvarez, MD, Principal Investigator — Divison of Gynecologic Oncology at University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States